CLINICAL TRIAL: NCT02552329
Title: A Randomized Controlled Trial of Mind-body Exercise: Effects of a 6-month Tai Chi Exercise on Cognition and Serum Biomarkers of Individuals With Mild Cognitive Impairment (MCI)
Brief Title: Effects of Tai Chi Exercise on Cognition and Serum Biomarkers of Individuals With MCI
Acronym: MCI-TaiChi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Somporn Sungkarat, associate professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chiang Mai University
Record Dates: First submitted 2014-01-16; First posted 2015-09-17 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; Tai Chi; cognitive functions
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Since no medication or other treatments are currently approved by Food and Drug Administration (FDA) for treatment of MCI, participants in the usual care group will not receive any form of treatment. They will receive an educational material about cognitive impairment. They will also be asked to maintain their daily routine.
- Tai Chi exercise group (Experimental): The Tai Chi exercise group will exercise for 50 minutes/session, 3 times /week for 24 consecutive weeks (6 months). Each 50-minute session will include a 10-minute warm up, 30-min exercise, and 10-min cool down.
  Interventions: Other: Tai Chi exercise

INTERVENTIONS:
Other: Tai Chi exercise — The Tai Chi exercise group will exercise for 50 minutes/session, 3 times /week for 24 consecutive weeks (6 months). Each 50-minute session will include a 10-minute warm up, 30-min exercise, and 10-min cool down, The 10 forms Tai Chi will be used.
  Arms: Tai Chi exercise group

SUMMARY:
Most research on Tai Chi has been done in the area of balance and falls. Studies examining the effects of Tai Chi exercise on cognitive function are sparse especially in the population of MCI. Therefore, the aims of the present study are: 1) to examine the effects of Tai Chi exercise on cognitive function of elderly with MCI, and 2) to investigate the effects of 6-month Tai Chi exercise on serum biomarkers in individuals with MCI.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) is a transitional stage before converting from normal aging to dementia. Older adults with MCI are 10 times more likely to develop dementia than cognitively intact older adults. Thus, strategies that could deter the conversion from MCI to dementia will have significant impact on public health.

There is growing interest in non-pharmacological approaches that could potentially slow down cognitive decline in late life. One such approach is the use of exercise to improve cognitive function. There is substantial evidence that exercise has benefits for cognitive function in elderly persons. Evidence on the benefits of exercise for cognition (either cognitive improvement or reduced cognitive decline) has been demonstrated through epidemiological studies, meta-analytical studies, and randomized controlled trials.

Although exercise training holds promise for delaying the onset and slowing down the progression of cognitive impairment among elderly persons, most studies utilized aerobic-base exercise with relatively high intensity. High intensity aerobic exercise may not be practical for older people because they are likely to have physical limitations and/or co-morbid diseases.Thus, the effects of other forms of exercise particularly those that are less intense and well suited to elderly conditions should be examined. The moderating factors linking exercise training and cognitive improvement is yet to be further investigated.

Tai Chi, a form of mind-body exercise, is a popular exercise among elderly. Although Tai Chi is considered as an aerobic exercise, the focus of this exercise in elders is not on cardiovascular fitness. It is characterized by slow, gentle motion and emphasized the conscious control of body movements. Several cognitive components including attention and mindfulness engage with physical movements during Tai Chi exercise. Thus, it is expected that Tai Chi exercise would have great benefit on cognition. Most research on Tai Chi has been done in the area of balance and falls. Studies examining the effects of Tai Chi exercise on cognitive function are sparse especially in the population of mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis for MCI based on Petersen's criteria as follows:

   * A self-reported memory complaint, corroborated by an informant interview
   * A score on a standardized memory test rated as 0.5 on Clinical Dementia Rating (CDR)
   * Normal general cognitive function, as determined by a clinician's judgment based on a structured interview with the patient and an informant report and adjusted Thai Mini-Mental State Examination (TMSE) 35
   * No or minimal impairment in activities of daily living (ADLs) or instrumental Activity of Daily Living (IADL), as determined by clinical review with the patients and informant interview
   * Not sufficiently impaired, cognitively and functionally, to meet National Institute of Neurological and Communicative Disorders and Stroke/ Alzheimer's disease and Related Association (NINCDS-ADRDA) criteria for AD, as judged by an experienced AD clinician
2. Presence of cognitive impairment determined by the score on the Montreal Cognitive Assessment (MoCA) lesser than 26
3. Comprehend instructions and willing to participate

Exclusion Criteria:

1. Presence of medical conditions that would be unsafe to exercise
2. Presence of neurological conditions (e.g. Parkinson's disease, Stroke, Multiple Sclerosis)
3. Presence of depressive symptoms, defined by the Geriatric Depression Scale (GDS)-Thai version 36
4. Presence of acute or/and chronic disease that could not be controlled (e.g. Arthritis, Asthma, Hypertension, Diabetes mellitus, Coronary artery disease)
5. Taking alcohol 6 hr before testing or using drug regimens that affect performance such as sedative and antidepressant.
6. Exercise regularly (40-50 min/day at least 3 days/week)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cognitive functions at 6 months | 6 months
  memory, attention, executive function will be evaluated

SECONDARY OUTCOMES:
Change from baseline in serum biomarkers at 6 months | 6 month
  inflammatory markers will be evaluated.
Change from baseline in fall risk at 6 months | 6 months
  Fall risk index will be evaluated using physiological profile approach (PPA)
Change from baseline in quality of life at 6 months | 6 months
  Health related quality of life will be evaluated using the Short Form 36 (SF-36) questionnaire.
Change from baseline in cognitive functions at 3 months | 3 months
  memory, attention, executive function will be evaluated
Change from baseline in fall risk at 3 months | 3 months
  Fall risk index will be evaluated using physiological profile approach (PPA)

CONTACTS AND LOCATIONS:
Overall Officials: Somporn Sungkarat, PhD, Principal Investigator — Department of Physical Therapy, Faculty of Associated Medical Sciences, Chiang Mai, Thailand
Locations (1):
- Department of Physical Therapy, Faculty of Associated Medical Sciences, Chiang Mai University, Maung, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No